CLINICAL TRIAL: NCT01173367
Title: Assessment of the Safety of Anti-pyretic Therapy in Critically Ill Adults
Brief Title: Anti-pyretic Therapy in Critically Ill Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Intensive Care Foundation (Other)
Responsible Party: Principal Investigator, Daniel Niven, Intensivist, Department of Critical Care Medicine, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-23090
Record Dates: First submitted 2010-07-28; First posted 2010-08-02 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Fever
Keywords: Fever; ICU; Acetaminophen; Inflammatory mediators; Safety
MeSH Terms: conditions — Fever

ARMS (2):
- Aggressive Fever Treatment (Active Comparator)
  Interventions: Other: Aggressive Fever Treatment
- Permissive Fever Treatment (Active Comparator)
  Interventions: Other: Permissive Fever Treatment

INTERVENTIONS:
Other: Aggressive Fever Treatment — Patients assigned to the aggressive fever treatment protocol will receive acetaminophen 650 mg enterally every 6 hours for fever ≥ 38.3°C and external cooling will be initiated for temperatures ≥ 39.5°C. Acetaminophen and external cooling will be discontinued once core temperature is less than 38.3°C and 39.5°C respectively.
  Arms: Aggressive Fever Treatment
Other: Permissive Fever Treatment — Patients assigned to the permissive treatment strategy will not receive anti-pyretic therapy until the temperature reaches 40.0°C at which point they will receive acetaminophen 650mg every 6 hours. External cooling will be initiated for temperatures ≥ 40.5°C. Acetaminophen and external cooling will be discontinued once core temperature is less than 40.0°C and 40.5°C respectively.
  Arms: Permissive Fever Treatment

SUMMARY:
The impact of fever and its management in different medical and surgical populations of critically ill patients has not been explained to date. The current study aims to assess the safety and efficacy of treatment of critically ill patients with a permissive versus aggressive fever treatment strategy.

DETAILED DESCRIPTION:
The impact of fever and its management in different medical and surgical populations of critically ill patients has not been explained to date. Clinical trials in critically ill surgical patients have demonstrated null or potentially harmful effects of treatment of moderate degrees of fever. However, the pathophysiological effects of fever treatment are not well defined according to different patient populations, and clinical trial results are questionably generalized to medical ICU patients. This may relate to different mechanisms of fever in these populations and merits further investigation. There is also very little known about the exact timing of expression of the diverse pro and anti-inflammatory mediators involved in inducing, maintaining and eventually abrogating the fever response. Treating on the sole basis of an elevated temperature may lead to detrimental effects if the anti-inflammatory cascade naturally regulating this response is active, demonstrating the importance of understanding the normal pattern of regulation of these diverse mediators. The current study aims to assess the safety and efficacy of treatment of critically ill patients with a permissive versus aggressive fever treatment strategy. In addition, the effect of anti-pyretic therapy on markers of inflammation in neurologically intact critically ill adults will be evaluated.

The study population will be neurologically intact febrile adults (≥18 years) admitted to the Peter Lougheed Center (PLC) or Foothills Medical Center (FMC) ICU over a 12-month period in Calgary, Alberta, Canada. Consenting patients that fulfill enrolment criteria will be randomly allocated to either the permissive or aggressive treatment group (see Interventions section for details). Randomization will be concealed using the consecutively numbered sealed opaque envelope technique. Samples of blood will be collected from study patients at enrolment and subsequently at 12, 24 and 48 hours for assessment of inflammatory mediators.

Markers of feasibility will include the rate of enrolment, adherence of patients to assigned treatment regimen/protocol violation, acceptance of the protocol by staff, and facility and maintenance of random allocation technique. Markers of safety will include potential adverse events such as 28-day survival, nosocomial infection rate, and evidence of myocardial ischemia, or hepatocellular inflammation during the febrile episode.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Fever (two consecutive measurements ≥ 38.3°C at least 2 hours apart or a single temperature measurement ≥ 39.5°C)
* Admitted to ICU with an expected length of stay at least 48 hours related to critical illness
* Attending physician approval

Exclusion Criteria:

* Admission to ICU for support for specific procedure (e.g. endoscopy, acute dialysis, bronchoscopy)
* Acute brain injury due to any etiology
* Acute myocardial ischemia
* Documented hepatitis with elevated alanine aminotransferase (ALT) more than twice the upper limit of normal, or chronic hepatic failure (defined by evidence of cirrhosis on available imaging or known varices, ascites, hepatic encephalopathy, hepatorenal syndrome, and/or hepatocellular carcinoma)
* Hyperthermia syndromes (malignant hyperthermia, heat stroke, neuroleptic malignant syndrome, serotonin syndrome, or endocrine causes including thyrotoxicosis, pheochromocytoma, and adrenal crisis)
* Refractory shock with lactic acidosis >4 mmol/L (at the time of screening for study enrollment) despite supportive therapy or need for paralytic treatment to reduce metabolic demand
* Requirement for use of anti-pyretic agents (acetaminophen or NSAIDs) for indications other than treatment of fever
* Receipt of anti-pyretic pharmacotherapy within 6-hours of expected study enrollment (650mg acetaminophen, 800mg ibuprofen, or 325mg acetylsalicylic acid)
* Contraindications to esophageal temperature monitoring
* Pregnancy (all women of child-bearing potential need to have a pregnancy test performed prior to enrollment)
* Time from onset of fever in the ICU to consideration for study enrollment is > 12 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
28-day survival | 28-day

SECONDARY OUTCOMES:
Feasibility of randomizing critically ill patients to different fever management strategies | 12 months
Consumption of anti-microbials | Maximum 28-days from enrollment
Incidence of nosocomial infection | Maximum 28-days from enrollment
The effect of anti-pyretic treatment of fever on markers of inflammation | 48 hours
Incidence of myocardial infarction during treatment of fever | Maximum 28-days from enrollment
Incidence of hepatocellular inflammation related to acetaminophen use | Maximum 28-days from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Laupland, MD MSc FRCPC, Principal Investigator — Faculty of Medicine, University of Calgary; Henry T Stelfox, MD PhD FRCPC, Principal Investigator — Faculty of Medicine, University of Calgary
Locations (2):
- Canada (2):
  - Intensive Care Unit, Peter Lougheed Center, Calgary, Alberta
  - Intensive Care Unit, Foothills Medical Center, Calgary, Alberta

REFERENCES:
- [Derived] Niven DJ, Stelfox HT, Leger C, Kubes P, Laupland KB. Assessment of the safety and feasibility of administering antipyretic therapy in critically ill adults: a pilot randomized clinical trial. J Crit Care. 2013 Jun;28(3):296-302. doi: 10.1016/j.jcrc.2012.08.015. Epub 2012 Oct 24. PMID 23102531
- [Derived] Niven DJ, Leger C, Kubes P, Stelfox HT, Laupland KB. Assessment of the safety and feasibility of administering anti-pyretic therapy in critically ill adults: study protocol of a randomized trial. BMC Res Notes. 2012 Mar 16;5:147. doi: 10.1186/1756-0500-5-147. PMID 22420838